CLINICAL TRIAL: NCT02948439
Title: Exercise and Neurovascular Function During Pregnancy
Brief Title: Prenatal Exercise and Cardiovascular Health (PEACH)
Acronym: PEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00061045
Record Dates: First submitted 2016-07-13; First posted 2016-10-28 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy
Keywords: pregnancy; cardiovascular; nervous system; exercise
MeSH Terms: conditions — Neurologic Manifestations; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention (Experimental): The aerobic exercise intervention will consist of a walking program at 50-70% of individual heart rate reserve. This will begin at 16-20 weeks gestation and continue 3-4 times per week until the end of the study (34-36 weeks). The duration of exercise will increase each week up to a maximum of 40 minutes (5 min warm up, 25 minutes exercise, 5 min cool down). Women will have at least one supervised exercise session per week. The investigators will also monitor other activity using questionnaires and accelerometry. This will occur at baseline (16-20 weeks), mid-intervention (24-26 weeks) and at the end (34-36 weeks).
  Interventions: Other: Aerobic exercise
- Control Group (No Intervention): These women will continue regular daily activities. Activity will be monitored periodically with questionnaires and accelerometry. This will occur at baseline (16-20 weeks), mid-intervention (24-26 weeks) and at the end (34-36 weeks).

INTERVENTIONS:
Other: Aerobic exercise — Brisk walking 3-4 times per week for up to 40 minutes of activity.
  Other Names: walking program
  Arms: Exercise Intervention

SUMMARY:
Maintenance of a healthy pregnancy depends on an appropriate adaptation and responsiveness of blood vessels, to ensure appropriate blood flow to the fetus during everyday stressors. Previous work by the investigators has demonstrated that during pregnancy, the part of the nervous system responsible for cardiovascular function (the sympathetic nervous system) is hyperactive. The investigators also know that in women who develop high blood pressure during pregnancy that sympathetic nervous system activity is even higher. Yet, very little is known about why this occurs and how this might be affected.

Pregnant women are encouraged to be active, yet, less than 15% of women perform sufficient exercise to meet current guidelines. This is important because hyperactivity of the sympathetic nervous system is observed in other inactive populations and has been linked to adverse cardiovascular health outcomes including hypertension, atherosclerosis, heart attack, and stroke. Indeed, in 2011, the American Heart Association stated that inactivity was a risk factor as potent as cigarette smoking for the development of future cardiovascular disease in women.

The investigators' work and others have demonstrated that exercise during pregnancy is beneficial for both the mom and baby; however, the effect of prenatal exercise on neurovascular function is not known. If exercise is effective in controlling the increase in sympathetic activity that occurs during pregnancy, or its effects on the cardiovascular system, this may help prevent the development of high blood pressure or other cardiovascular problems during pregnancy.

DETAILED DESCRIPTION:
The objectives of this study are to: 1) examine the impact of exercise on sympathetic and vascular function during pregnancy; 2) examine the role of endothelial function on the vascular effects of exercise during pregnancy.

Study design:

100 women (>18yrs) will be recruited in the first or second trimester (<20 wks). Women with multiple pregnancies will be excluded. Eligible women will be randomized between an aerobic exercise intervention (EXER) or no intervention (CTRL).

Initial testing will take place between 16-20 weeks of pregnancy. Following initial baseline testing, women will be randomly assigned to an exercise intervention or no intervention. Women will receive an opaque sequentially numbered envelop with their allocation. Allocation will be determined using a randomly generated allocation sequence by an individual not associated with the research study. The intervention will consist of aerobic exercise equivalent to 50-70% of heart rate reserve, 3-4 times per week until the end of the study (34-36 weeks). For initial baseline testing (16-20 weeks) and at the end of the intervention (34-36 weeks), participants will visit the laboratory twice

On Day 1, participants will complete a peak exercise test on the treadmill or bike to volitional fatigue to measures fitness and cardiovascular/cerebrovascular responses to exercise.

On Day 2 Participants will arrive fasted (12 hrs) and blood samples will be collected. Anthropometrics, personal/familial history of hypertension and pregnancy complications will be recorded. Following a standardized breakfast, participants will undergo an assessment of reflex neurovascular control including a cold pressor test, flow mediated dilation and end expiratory voluntary breath hold. Muscle sympathetic nerve activity, ultrasound (blood flow and diameter of brachial, femoral and carotid arteries), blood pressure, heart rate and respiratory variables will be measured.

OUTCOME/IMPACT

Pregnancy is a stress-test for life; with women who develop complications during pregnancy having a higher risk for cardiovascular disease later in life. Exercise is well known to prevent cardiovascular disease through improvements in endothelial function and the sympathetic nervous system. Whether this improvements is also seen in pregnancy remains to be seen.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* singleton pregnancy
* cleared to exercise by health care provider using Par Med X for Pregnancy (CSEP)

Exclusion Criteria:

* multiple gestation
* absolute contraindication to exercise (CSEP)
* <18 years old
* develops any contraindication during intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Sympathetic Nerve Activity - cold pressor test response | 16-20 weeks and 34-36 weeks gestation
  Response of the sympathetic nervous system to cold pressor test (% change in activity)

SECONDARY OUTCOMES:
Respiratory measures - respiratory frequency | 16-20 weeks and 34-36 weeks gestation
  Breathing frequency (breaths per minute). Measured using spirometry.
Sympathetic Nerve Activity - breath hold response | 16-20 weeks and 34-36 weeks gestation
  Response of the sympathetic nervous system to voluntary breath hold (% change in activity)
Respiratory measures - tidal volume | 16-20 weeks and 34-36 weeks gestation
  Tidal Volume (Liters per breath). Measured using spirometry.
Respiratory measures - oxygen | 16-20 weeks and 34-36 weeks gestation
  Oxygen metabolism (% oxygen used per breath). Measured using a gas analyzer.
Respiratory measures - carbon dioxide | 16-20 weeks and 34-36 weeks gestation
  Carbon Dioxide production (% carbon dioxide per breath). Measured using a gas analyzer.
Respiratory measures - lung volume | 16-20 weeks and 34-36 weeks gestation
  Total Lung Capacity (Liters). Measured using spirometry.
Cerebral blood flow at rest | 16-20 weeks and 34-36 weeks gestation
  Brain blood flow in the middle cerebral artery at rest (cm/s). Measured using transcranial doppler ultrasound.
Cerebral autoregulation | 16-20 weeks and 34-36 weeks gestation
  Brain blood flow in the middle cerebral artery in response to standing (cm/s). Measured using transcranial doppler ultrasound.
Cerebral blood flow during exercise | 16-20 weeks and 34-36 weeks gestation
  Brain blood flow in the middle cerebral artery during the acute incremental peak exercise test (cm/s). Measured using transcranial doppler ultrasound.
fasted blood sample - blood volume | 16-20 weeks and 34-36 weeks gestation
  Fasted blood samples (~30ml) will be analyzed for markers of blood volume (hematocrit; %)
fasted blood sample - neurotransmitters | 16-20 weeks and 34-36 weeks gestation
  Fasted blood samples (~30ml) will be analyzed for sympathetic nervous system neurotransmitters (Norepinephrine, Epinephrine, Neuropeptide-Y).
fasted blood sample- inflammatory markers | 16-20 weeks and 34-36 weeks gestation
  Fasted blood samples (~30ml) will be analyzed for inflammatory markers (i.e. C-Reactive Protein).
fasted blood sample- epigenetics | 16-20 weeks and 34-36 weeks gestation
  Fasted blood samples (~30ml) will be analyzed for epigenetics (optional).
fasted blood sample- sex hormones | 16-20 weeks and 34-36 weeks gestation
  Fasted blood samples (~30ml) will be analyzed for sex hormones (estrogen, progesterone, testosterone).
fasted blood sample- metabolic | 16-20 weeks and 34-36 weeks gestation
  Fasted blood samples (~30ml) will be analyzed for metabolic parameters (i.e. glucose)
fetal outcomes- birth weight | within one month postpartum
  Participants will provide the investigators with birth weight for the infant (grams).
fetal outcomes- length | within one month postpartum
  Participants will provide the investigators with birth length for the infant (cm).
fetal outcomes- gestational age | within one month postpartum
  Participants will provide the investigators with gestational age at delivery (weeks).
maternal outcomes- mode of delivery | within one month postpartum
  Participants will provide the investigators with mode of delivery (vaginal or cesarean).
maternal outcomes- delivery complications | within one month postpartum
  Participants will provide the investigators with information regarding any delivery complications.
maternal outcomes- pregnancy complications | any time during study
  Participants will provide the investigators with information regarding any pregnancy complications (gestational diabetes, pregnancy induced hypertension, preeclampsia).
fetal outcomes- apgar score | within one month postpartum
  Participants will provide the investigators with APGAR scores (out of 10) for the infant
fetal outcomes- NICU | within one month postpartum
  Participants will provide the investigators with information regarding length (days) of admission to Neonatal Intensive Care Unit (NICU) if applicable.
maternal outcomes- gestational weight gain | within one month postpartum
  Participants will provide the investigators with the last maternal weight immediately before delivery. This will be used to calculate gestational weight gain (kg; last maternal weight - self reported pre-pregnancy weight).
Endothelial Function - time to peak dilation | 16-20 weeks and 34-36 weeks gestation
  The investigators will assess endothelial function using flow mediated dilation (FMD, time to maximal dilation; s)
Endothelial Function- flow mediated dilation | 16-20 weeks and 34-36 weeks gestation
  The investigators will assess endothelial function using flow mediated dilation (change in diameter; mm)
Endothelial Function - shear stress | 16-20 weeks and 34-36 weeks gestation
  The investigators will assess endothelial function using flow mediated dilation (shear stress; pascals).
Accelerometry | 16-20 weeks and 34-36 weeks gestation
  The investigators will objectively measure physical activity using an accelerometer for one week. Average number of minutes per day spent in various activity levels will be determined.
Physical Activity Questionnaire | 16-20 weeks and 34-36 weeks gestation
  The participants will report physical activity using the pregnancy physical activity questionnaire (gives metabolic equivalent hours per week (MET-hr/week).
Depression rating | 16-20 weeks and 34-36 weeks gestation
  Participants will answer a 10-question questionnaire regarding their mood. A score of 10 or higher is indicative of depressive symptoms. The investigators will report the over number of women in each group who have a score of 10+ at the start and end of the intervention.
Sleep Quality | 16-20 weeks and 34-36 weeks gestation
  Participants will report their sleep quality using the Pittsburgh Sleep Quality index. A score of 5 or more indicates poor sleep quality. The investigators will compare this score between groups before and after the intervention.
Food log | 16-20 weeks and 34-36 weeks gestation
  The investigators will objectively measure nutrients in diet using a three day food record. This is completed through Food Prodigy/ Food Processor software.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Skow, MSc, Study Director — University of Alberta
Locations (1):
- Program for Pregnancy and Postpartum Health, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boparai R, Skow RJ, Farooq S, Steinback CD, Davenport MH. Prenatal exercise and cardiovascular health (PEACH) study: the remote effect of aerobic exercise training on conduit artery and resistance vessel function. Appl Physiol Nutr Metab. 2021 Dec;46(12):1459-1468. doi: 10.1139/apnm-2020-0902. Epub 2021 Jun 23. PMID 34161737
- [Derived] Skow RJ, Fraser GM, Steinback CD, Davenport MH. Prenatal Exercise and Cardiovascular Health (PEACH) Study: Impact on Muscle Sympathetic Nerve (Re)Activity. Med Sci Sports Exerc. 2021 Jun 1;53(6):1101-1113. doi: 10.1249/MSS.0000000000002583. PMID 33315812

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT02948439/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT02948439/ICF_001.pdf